CLINICAL TRIAL: NCT02700035
Title: A Randomized Control Trial (RCT) of a Family-Centered Ojibwe Substance Abuse Prevention
Brief Title: A Family-Centered Ojibwe Substance Abuse Prevention
Acronym: BZDDD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nebraska Lincoln (Other)
Collaborators: Johns Hopkins University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 14158
Record Dates: First submitted 2016-02-26; First posted 2016-03-07 (Estimated); Last update posted 2022-03-11 (Actual); Status verified 2022-03

CONDITIONS: Substance Use
Keywords: Intervention; Prevention; Randomized Controlled Trial; Bii-Zin-Da-De-Dah
MeSH Terms: conditions — Substance-Related Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- BZDDD Prevention Program Intervention (Experimental): We employed an experimental randomized block (RB) design; blocked on reservation where 157 were assigned to the intervention condition (Bii-Zin-Da-De-Dah (Listening to One Another) 14 week family based prevention program). The first 4 weeks of the program are oriented towards the Anishinabe cultural traditions and the traditional Anishinabe family. Weeks 5 through 8 focus on identifying feelings and how to manage negative feelings such as anger and sadness in positive ways. The last 6 weeks of the program focus on outside influences and how to build positive support systems. Prior to the intervention, we completed a pre-test with families in the experimental group. Following the program, we completed a post-test and a 6-month youth follow-up.
  Interventions: Other: Bii-Zin-Da-De-Dah (Listening to One Another)
- BZDDD Prevention Program Control (No Intervention): We employed a randomized block (RB) design; blocked on reservation, 147 families were randomly assigned to the control condition. We completed a post-test and a 6-month youth follow-up.

INTERVENTIONS:
Other: Bii-Zin-Da-De-Dah (Listening to One Another) — Bii-Zin-Da-De-Dah (Listening to One Another) is a family-centered alcohol and drug prevention program for Anishinabe communities. It was the first American Indian adaptation of the Iowa Strengthening Families Program (now called the Strengthening Families Program). This program has been developed and adapted in partnership with multiple Anishinabe communities over a span of 13 years. Bii-Zin-Da-De-Dah has been enormously popular in communities. It is currently the center piece of a National Canadian Mental Health Promotion Program funded by the Public Health Agency of Canada. Now in its third Phase, focusing on national scale-up among first nations people, it has been adapted for eight cultures and translated into French in a recent implementation in Canada.
  Other Names: BZDDD
  Arms: BZDDD Prevention Program Intervention

SUMMARY:
This study will complete a multisite randomized controlled trial (RCT) of a family-centered alcohol and drug prevention program for Anishinabe (Ojibwe) pre-adolescents in 3rd or 4th grade (Fall 2017) or who are age 8-10 years on June 1, 2017. The 14 week program includes cultural lessons to strengthen family interactions, decrease substance use, teach parenting skills, increase social skills, improve refusal skills, and teach coping mechanisms for adolescents and parents. Session are expected to last around 3-hours, including a meal, youth and parent breakout sessions, and group based discussions. Parents and adolescents will participate in a pre-test before the program begins and a series of post-tests after the program ends.

DETAILED DESCRIPTION:
Investigators will implement a multisite randomized controlled trial (RCT) of a family-centered alcohol and drug prevention program for Anishinabe (Ojibwe) pre-adolescents in 3rd or 4th grade (Fall 2017) or who are age 8-10 years on June 1, 2017. to assess its efficacy for delaying and/or preventing adolescent onset of alcohol and drug use. This unique project will empirically address cultural challenges for RCTs involving AI cultures by evaluating contamination and informal diffusion in AI communities and extended families. AI values of sharing and community benefits clash with Western RCT methods of withholding benefits from control groups vs. treatment groups. Although risks of informal community dissemination and control group contamination are widely acknowledged challenges for AI RCTs, the degree to which this actually occurs and the potential impact has never been assessed. Rather, efforts are made to suppress and minimize AI values that result in informal dissemination and contamination, or the potential effects are simply ignored. This research will address these challenges by attempting to measure and control for them. The intent-to-treat study design will allow us to use question routing aimed at identifying content sharing among treatment and control adolescents and their treatment and control group parents. Moreover, the project will also use question routes to investigate potential contamination via extended family members who have contact with both the treatment and control families. Investigators will then assess potential impact of measured contamination on observed intervention effects.

At the completion of the study, Investigators will work with community research partners to develop a plan to sustain the prevention program. A sustainability plan is part of our model for developing and implementing culturally specific evidence-based prevention programs. Communities have readiness for sustainability due to familiarity and the popularity of BZDDD. We will work through community advisory boards (named Prevention Research Councils or PRCs) to place the program within schools, health services, and social services agencies. The project will leave behind comprehensive facilitator manuals in addition to a videotaped training program to facilitate ongoing training. In addition, the program has recently been adapted to a virtual program in response to COVID-19. The investigative team has a proven track record of sustainability in prior adaptions of BZDDD.

ELIGIBILITY:
Inclusion Criteria:

* Youth who self-Identified as American Indian (between the ages of 8-10)
* Adult Guardians of participating youth (aged 18 or older)

Exclusion Criteria:

* Youth who did not self-identify as American Indian
* Youth under the age of 8 years old
* Youth over the age of 11 years old.

Ages: 8 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 705 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2020-11 (Actual); Study Completion 2020-11 (Actual)

PRIMARY OUTCOMES:
Change in Cigarette Use | Pre-Test Baseline, 15 Week, 6 Month
  Frequency of use of cigarettes
Change in Alcohol Use | Pre-Test Baseline, 15 Week, 6 Month
  Frequency of use of alcohol
Change in Illicit Drug Use | Pre-Test Baseline, 15 Week, 6 Month
  Frequency of use of illicit drug use

CONTACTS AND LOCATIONS:
Overall Officials: Leslie B Whitbeck, Ph.D., Principal Investigator — University of Nebraska Lincoln

IPD SHARING:
Plan to Share IPD: No
Due to the nature of the collaboration with tribal entities, the data will not be made publicly available without approval of the collaborating tribal council government bodies.

REFERENCES:
- [Background] Whitbeck LB, Walls ML, Welch ML. Substance abuse prevention in American Indian and Alaska Native communities. Am J Drug Alcohol Abuse. 2012 Sep;38(5):428-35. doi: 10.3109/00952990.2012.695416. PMID 22931077
- [Background] Keogh-Brown MR, Bachmann MO, Shepstone L, Hewitt C, Howe A, Ramsay CR, Song F, Miles JN, Torgerson DJ, Miles S, Elbourne D, Harvey I, Campbell MJ. Contamination in trials of educational interventions. Health Technol Assess. 2007 Oct;11(43):iii, ix-107. doi: 10.3310/hta11430. PMID 17935683
- [Background] Lang DL, DiClemente RJ, Hardin JW, Crosby RA, Salazar LF, Hertzberg VS. Threats of cross-contamination on effects of a sexual risk reduction intervention: fact or fiction. Prev Sci. 2009 Sep;10(3):270-5. doi: 10.1007/s11121-009-0127-z. PMID 19241171
- [Background] Howe A, Keogh-Brown M, Miles S, Bachmann M. Expert consensus on contamination in educational trials elicited by a Delphi exercise. Med Educ. 2007 Feb;41(2):196-204. doi: 10.1111/j.1365-2929.2006.02674.x. PMID 17269954
- [Background] Spoth RL, Redmond C, Shin C. Reducing adolescents' aggressive and hostile behaviors: randomized trial effects of a brief family intervention 4 years past baseline. Arch Pediatr Adolesc Med. 2000 Dec;154(12):1248-57. doi: 10.1001/archpedi.154.12.1248. PMID 11115311
- [Background] Spoth RL, Redmond C, Shin C. Randomized trial of brief family interventions for general populations: adolescent substance use outcomes 4 years following baseline. J Consult Clin Psychol. 2001 Aug;69(4):627-42. doi: 10.1037//0022-006x.69.4.627. PMID 11550729
- [Background] Kosterman R, Hawkins JD, Haggerty KP, Spoth R, Redmond C. Preparing for the drug free years: session-specific effects of a universal parent-training intervention with rural families. J Drug Educ. 2001;31(1):47-68. doi: 10.2190/3KP9-V42V-V38L-6G0Y. PMID 11338965